CLINICAL TRIAL: NCT03296020
Title: The Efficacy of Honey on Improving the Post Surgical Course After Tonsillectomy in Children-prospective Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0079-17-EMC
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Honey

STUDY DESIGN:
Intervention Model Description: randomized clinical trials that included 2 armes: the control group and the case group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): After the surgery, during the hospitalization ,the control group would get as is customary in our ENT department :acetaminophen syrup+ syrup oxycode( as necessary).
  After the discharge from the hospital - the patients would take( as is customary in our ENT department): acetaminophen syrup ( as necessary) and other painkillers ( as necessary).
  The families would ask to follow treatment protocols for 7 days and will fill a questionnarie every day during the 7 days.
- case group-"HONEY" (Experimental): After the surgery, during the hospitalization ,the case group would instructed to use honey twice a day( 5 ml- one tea spoon each time)+acetaminophen syrup + syrup oxycode( as necessary).
  After the discharge from the hospital - the patients would take:acetaminophen syrup ( as necessary) and other painkillers+honey twice a day( 5 ml- one tea spoon each time) .
  The families would ask to follow treatment protocols for 7 days and will fill a questionnarie every day during the 7 days.
  Interventions: Other: HONEY

INTERVENTIONS:
Other: HONEY — 100% Natural pure Honey, produced by EIN HAROD CO-OPERATIVE, ISRAEL
  Arms: case group-"HONEY"

SUMMARY:
The aim of this study is to investigate the effect of honey administration on pain following pediatric tonsillectomy or adenotonsilectomy.

The patients( children 2-18 years old) will divide into two groups by simple randomization method( the control group and the case group).

After surgery the case group: would instructed to use honey twice a day( 5 ml- one tea spoon each time)+acetaminophen syrup+ syrup oxycode( as necessary).

the control group would get as is customary in our ENT department :acetaminophen syrup+ syrup oxycode( as necessary).

The families would ask to follow treatment protocols for 7 days. From the first to the 7th day after the operation , the parents would ask to fill a questionnaire every day for assessment of pain intensity by visual analouge scale(VAS) , the numbers of painkillers taken daily, the number of times the child awaking at night due to pain, the amount of fluids intake daily, the time of commencement of regular oral intake.

patient would follow up 7-14 days after surgery.

DETAILED DESCRIPTION:
This study was approved by the regional ethics committe of the Hospital. The participants would be: Children (2-18 years old, male and female), who will have the indication of tonsillectomy and will undergo classic tonsillectomy with or without adenoidectom in otolaryngology departement in HaEmek Hospital and they ate already honey in their lives.

Exclusion criteria:

* Allergy to honey
* Allergy to Acetaminophen
* Patients with Diabeties mellitus
* pregnent/breast feeding patients
* patients with coagulation disorders
* patients who undrego another operation in addition to tonsillectomy with or without adenoidectomy ( except insertion of ventilation tubes surgery).

ELIGIBILITY:
Inclusion Criteria:

* children ages 2-18 years old that candidates for Tonsillectomy with or without adenoidectomy surgery, in otolaryngolgy department , HaEmek Hospital, Afula.
* Parents' signature on informed consent form.

Exclusion Criteria:

* Allergy to honey
* Allergy to Acetaminophen
* Patients with Diabeties mellitus
* pregnent/breast feeding patients
* patients with coagulation disorders
* patients who undrego another operation in addition to tonsillectomy with or without adenoidectomy ( except insertion of ventilation tubes surgery).

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 7 days
  pain intensity by visual analouge scale(VAS), the numbers of painkillers taken daily, the number of times the child awaking at night due to pain
Amount of fluids | 7 days
  what is the amount of fluids intake daily
The time of commencement of regular oral intake. | 7-14 days
  How long is take post surgery for the child to return to his regular oral intake

CONTACTS AND LOCATIONS:
Overall Officials: tzvi chen, Study Chair — haemek medical center; tzvi chen, Study Director — haemek medical center; TZVI CHEN, Principal Investigator — haemek medical center
Locations (1):
- HaEmek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: Undecided